CLINICAL TRIAL: NCT04764890
Title: Effectiveness of Electro-acupuncture and Manual Therapy on Pain and Fucntion in Patients With Sciatica
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEUSPU12
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-02

CONDITIONS: Sciatica; Electroacupuncture; Manual Therapy
MeSH Terms: conditions — Sciatica | interventions — Electroacupuncture; Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Electroacupuncture and manual therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture and manual therapy (Experimental): Electroacupuncture in several points and manual therapy in the lumbar spine
  Interventions: Other: Electroacupuncture; Other: Manual therapy
- Manual therapy (Active Comparator): Manual therapy in the lumbar spina
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Electroacupuncture — Electroacupuncture in several point
  Arms: Electroacupuncture and manual therapy
Other: Manual therapy — Manual therapy in the lower spine.

SUMMARY:
The aims of the study are:

To study the pain efficacy of an electroacupuncture and manual therapy protocol versus the use of manual therapy in patients with sciatica.

To study the efficacy on function of an electroacupuncture and manual therapy protocol versus the use of manual therapy in patients with sciatica.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 50 years old.
* Diagnosis of sciatica

Exclusion Criteria:

* Pregnancy.
* Fear of needles.
* Coagulation disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-11 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale for pain | up to 5 weeks
  Pain measurement: 100-mm visual analog scale (VAS), horizontal line ranging from 0 mm (nopain) to 100 (worts imaginable pain)
Oswestry Low Back Pain Disability Questionnaire | up to 5 weeks
  This questionnaire has been designed to give us information as to how your back or leg pain is affecting your ability to manage in everyday life.

CONTACTS AND LOCATIONS:
Locations (1):
- CEU-San Pablo Universtiy, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided